CLINICAL TRIAL: NCT01963806
Title: Guided and Unguided CBT for Social Anxiety Disorder and/or Panic Disorder Via the Internet and a Smartphone Application
Brief Title: ACT-smart: Smartphone-supplemented iCBT for Social Phobia and/or Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Responsible Party: Principal Investigator, Per Carlbring, Professor, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT-smart
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Panic Disorder; Phobic Disorders
MeSH Terms: conditions — Panic Disorder; Phobic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Smartphone-supplemented iCBT with therapist support (Experimental): n = 50
  Interventions: Behavioral: Smartphone-supplemented iCBT; Behavioral: Therapist support
- Smartphone-supplemented iCBT without therapist support (Experimental): n = 50
  Interventions: Behavioral: Smartphone-supplemented iCBT
- Active waiting list control group with delayed treatment (Active Comparator): n = 50
  Interventions: Behavioral: Smartphone-supplemented iCBT; Other: Active waiting list

INTERVENTIONS:
Behavioral: Smartphone-supplemented iCBT — The Internet-administered cognitive behavioural self-help program (iCBT) will be divided into 10 weekly, progressively available modules covering CBT and Acceptance and Commitment Therapy (ACT) conceptualisations of anxiety disorders, as well as more specific therapeutic techniques such as cognitive restructuring, exposure training, attention and breathing exercises and relapse prevention . Each module also includes writing exercises.
  Also included is a tailored smartphone application. Briefly, the application allows the user to access, create and modify a personal database of behaviours and check-off these behaviours immediately when completed. Frequency of carried-out behaviours are recorded and displayed as statistics. The application also allows users to browse and search a database of behaviours uploaded by other study participants, providing both inspiration and a sense of social support.
Behavioral: Therapist support — The role of the therapists will be to provide feedback on the written exercises of each treatment module, as well as to provide support and encouragement. As a rule of thumb, the therapists will devote 15 minutes per participant and week.
  Arms: Smartphone-supplemented iCBT with therapist support
Other: Active waiting list — Completes measurements at day 24 and 48 and at the end of the initial treatment period, otherwise no activity until crossover.
  Arms: Active waiting list control group with delayed treatment

SUMMARY:
BACKGROUND: Smartphone technology presents a novel and promising opportunity to extend the reach of psychotherapeutic interventions by moving selected parts of the therapy into the real-life situations causing distress. This randomised controlled trial will investigate the effect of a transdiagnostic, Internet-administered cognitive behavioural (iCBT) self-help program for anxiety, supplemented with a tailored smartphone application. The effect of added therapist support will also be studied.

METHODS/DESIGN: 150 participants meeting diagnostic criteria for social anxiety disorder and/or panic disorder will be evenly randomised to one of three treatment arms: (1) smartphone-supplemented iCBT with therapist support; (2) smartphone-supplemented iCBT without therapist support; or (3) an active waiting list control group with delayed treatment. After the 10 week treatment period, the control group (3) will receive the same treatment as group (2). Primary outcome measure will be the Generalised Anxiety Disorder 7-item self-rating scale. Secondary measures include other anxiety, depression and quality of life measures. In addition to pre- and post-treatment measurements, the study includes two mid-treatment and two follow-up assessments (12 and 24 months).

HYPOTHESES: Based on prior research, we hypothesise that the therapist-guided form will be superior to the unguided form in reducing anxiety levels, and that both delivery modes will be superior to an active waiting-list control group.

ELIGIBILITY:
Inclusion Criteria:

* Satisfy DSM-IV-TR criteria for panic disorder and/or social anxiety disorder as assessed by the SCID.
* Daily access to the Internet via computer and smartphone
* Residing in Sweden and speaking sufficient Swedish to communicate with the research team

Exclusion Criteria:

* Parallel psychological treatment
* Non-stable dosage of psychoactive medication during last 3 months
* Participants deemed to suffer from suicidal tendencies or another condition requiring specialized treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The Generalised Anxiety Disorder 7-item (GAD-7) | Change from baseline at: [1] day 24 and [2] day 48 into the 10-week treatment period; [3] 0-1 week after the treatment period; follow-ups at [4] month 12 and [5] month 36 after the treatment period.
  The Generalised Anxiety Disorder 7-item (GAD-7). The 7 items of the scales are rated 0-3 ("Not at all" to "Nearly every day") based on their occurrence within the last 2 weeks. Good internal consistency and factor structure has been reported.

SECONDARY OUTCOMES:
Self-rated Liebowitz Social Anxiety Scale (LSAS-SR) | Change from baseline at: [1] 0-1 week after the treatment period; follow-ups at [2] month 12 and [3] month 36 after the treatment period.
Self-rated Panic Disorder Severity Scale (PDSS-SR) | Change from baseline at: [1] 0-1 week after the treatment period; follow-ups at [2] month 12 and [3] month 36 after the treatment period.
9-item Patient Health Questionnaire (PHQ-9) | Change from baseline at: [1] day 24 and [2] day 48 into the 10-week treatment period; [3] 0-1 week after the treatment period; follow-ups at [4] month 12 and [5] month 36 after the treatment period.
Quality of Life Inventory (QOLI) | Change from baseline at: [1] 0-1 week after the treatment period; follow-ups at [2] month 12 and [3] month 36 after the treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- Stockholm University, Stockholm, Sweden

REFERENCES:
- [Derived] Lindner P, Ivanova E, Ly KH, Andersson G, Carlbring P. Guided and unguided CBT for social anxiety disorder and/or panic disorder via the Internet and a smartphone application: study protocol for a randomised controlled trial. Trials. 2013 Dec 18;14:437. doi: 10.1186/1745-6215-14-437. PMID 24351088